CLINICAL TRIAL: NCT06601218
Title: A Phase I Study of the Effects of Cannabis on Cancer Burden: Placebo-Controlled, Double-Blind, Randomized Trial
Brief Title: Impact of Daily Oral Cannabis Doses in Patients With Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanna Babalonis, PhD (Other)
Responsible Party: Sponsor-Investigator, Shanna Babalonis, PhD, Associate Professor, College of Medicine, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 87078
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Cancer; Cancers, Pain
MeSH Terms: conditions — Neoplasms; Pain | interventions — Dronabinol

STUDY DESIGN:
Intervention Model Description: Randomization into 4 arms - each arm administers a dose of oral cannabis or placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1: Placebo Cannabis (Placebo Comparator): This arm will administer a placebo dose of oral cannabis (no active drug)
  Interventions: Drug: Placebo Comparator
- Arm 2: Active Cannabis Low (Active Comparator): This arm will administer an active low dose of cannabis
  Interventions: Drug: Oral cannabis low THC
- Arm 3: Active Cannabis High (Active Comparator): This arm will administer an active high dose of cannabis
  Interventions: Drug: Oral cannabis high THC
- Arm 4: Active Cannabis (THC+CBD) (Active Comparator): This arm will administer an active dose of cannabis (THC+CBD)
  Interventions: Drug: Oral cannabis THC/CBD

INTERVENTIONS:
Drug: Oral cannabis low THC — 4 months daily dosing with oral cannabis low THC
  Other Names: THC
  Arms: Arm 2: Active Cannabis Low
Drug: Placebo Comparator — 4 months of daily dosing with oral placebo
  Other Names: Placebo
  Arms: Arm 1: Placebo Cannabis
Drug: Oral cannabis high THC — 4 months of daily dosing with oral cannabis with high THC
  Other Names: THC
  Arms: Arm 3: Active Cannabis High
Drug: Oral cannabis THC/CBD — 4 months of daily dosing with oral cannabis with THC and CBD
  Other Names: THC/CBD
  Arms: Arm 4: Active Cannabis (THC+CBD)

SUMMARY:
This study will enroll patients with cancer and participants will be randomized to receive one dose of cannabis for approximately 4 months. There is a 3/4 (or 75%) chance that a participant will receive an active cannabis dose in the study. There is a 1/4 (or 25% chance) that a participant will receive a placebo dose (meaning a blank dose/no cannabis/no active drug). The goals of this study are to determine 1) the safety and tolerability of cannabis in individuals with cancer and 2) if cannabis can help with the side effects of cancer and cancer treatment - including nausea and vomiting, appetite, pain, sleep, and quality of life.

DETAILED DESCRIPTION:
Primary Objective: To evaluate the safety and tolerability of daily oral cannabis administration (5 mg THC, 15 mg THC, 15 mg THC+15 mg CBD) relative to placebo in patients with cancer who are on an active anti-cancer therapy. The percent of patients who elect to withdrawal from the study or removed by physician/investigators due AEs or safety concerns in each group will be measured and compared to the placebo group.

Secondary Objectives:

1. To evaluate frequency and severity of safety criteria violations from dosing to 4 hrs post-dose (HR, O2 saturation from fitness tracker).
2. To evaluate the percent of patients who withdrawal from the study or removed by physician/investigators for all reasons.
3. To determine final tolerated dose for future study (investigator determination after review of AEs, participant rated VAS, vitals).
4. To evaluate the effects of cannabis on cancer burden total score, as measured by the NCCN/Functional Assessment of Cancer Therapy (FACT) Symptom Index, a validated questionnaire that assesses cancer burden in the form of symptoms and concerns. Specifically, 17 items form 4 subscales that assess Disease-Related Symptoms-Physical (DRS-P), Disease- Related Symptoms-Emotional (DRS-E), Treatment Side Effects (TSE), and Function/Well-Being (F/WB). A total score is generated and will be assessed at baseline, during experimental dosing and follow-up.

Participants: Participants will be adult cancer patients, ages 18 and older, who have a histologically or cytologically confirmed locally advanced or metastatic solid tumor. These patients will be actively undergoing anti-cancer therapy, having been on a current regimen for at least one month prior to enrollment. An ECOG performance status of ≤2 and adequate organ and marrow function at baseline is required. A total of 80 patients will be enrolled in this study (n=20/arm).

Investigators will recruit participants from the University of Kentucky Markey Cancer Center. Patients who appear to meet basic/initial study criteria will be approached by Dr. and Doctor's team. Investigators will provide the patient with a study information card that contains basic information about the study and the contact information (e.g., phone, text, email, social media contacts) for the UK Center on Drug and Alcohol Research (CDAR; Dr. Babalonis and her team). When contacting the CDAR, the participant will have a chance to speak to staff and ask questions and will also have the opportunity to schedule an in-person screening appointment (the first of two in-person screening appointments).

Study Design: This study will utilize a randomized, double-blind, placebo-controlled, 4 arm design (n=80, n=20/arm). The study duration will be approximately 5.5 months, including 2 weeks of baseline (no drug administered), 4 months of daily dosing (including approx. 2 weeks of dose titration at the beginning of dosing, 3 months at target dose, approx. 2 weeks dose taper at the end of dosing), and a 1-month follow-up period (no drug administered).

All study participants will be randomized 1:1:1:1 by the study statistician, Dr. Donglin Yan. All patients are allowed to continue with anti-cancer therapies (but not cannabinoid-based medications) while enrolled in this study. Patients taking checkpoint inhibitors or with HPV-positive cancers will not be enrolled due to evidence (albeit limited) that concomitant cannabis reduces the efficacy of checkpoint inhibitors.

After enrollment and a minimum of a 2-week period of baseline data collection, a participant will begin receiving experimental cannabis/matched placebo doses. Investigators plan to administer one blinded dose per day during the approx. 4-month dosing protocol (including titration and taper). One oral (i.e., edible) daily dose will be administered on an outpatient basis. Due to DEA regulations (e.g., cannabis is a Schedule I drug with many regulatory restrictions), a trained research staff will visit the participant home approx. once per week to deliver approx. 1-2 week supply of doses. Each dose will be locked in its own safe and each safe will have a unique combination code (with an AirTag embedded in the safe for dose tracking capabilities if needed).

Participants will FaceTime or video chat with a research team member (at a pre-specified time) every day. During this video call, the participant will be provided a code to unlock one safe. The research staff member will ask the participant to open the safe and show the dose and its label on camera. The research staff will verify the correct participant name, date and dose code.

During this call, the research staff will also remind the participant to wear the fitness tracker per protocol so that the study team can monitor vitals (HR, O2) prior to and for 4 hrs post-dose. Participants will also be provided instructions to call the on-call physician/RN if not feeling well or if an alarm on the fitness tracker is received. The participant will be required to consume the dose on camera. This rationale for verification of dosing is three-fold: 1) to ensure no diversion occurs (i.e., the dose is consumed by the patient and not diverted to another person), 2) to verify study dosing adherence and 3) to ensure that the correct dose was administered (particularly early and late in the study when doses will be titrated and tapered). Participants are compensated for compliance with these calls.

If a participant has known travel, investigators will discuss the travel plans to determine if it is safe and advisable to take doses with them (in most scenarios, travel with doses will not be likely, but this will be discussed at the time of consent and when travel arises). In these scenarios, or at other times the participant is unavailable (e.g., hospitalized), the investigators/study physician will discuss a plan (e.g., not delivering scheduled doses, picking up unused doses, re-starting a titration schedule if a long break is anticipated, discharging from the study as a last resort).

Daily assessments for this study include video calls and app-based questionnaires. Participants will complete brief daily questionnaires via a smartphone app, covering morning assessments of sleep quality, hot flashes, night sweats, appetite, nausea, pain, and overall mood, as well as post-dose assessments of drug effects, mood, and vitals.

The in-home visits by a research assistant or nurse will include dose drop-off, review of adverse events, and addressing any study-related concerns. Monthly in-laboratory visits will assess adverse events, study progress, and continued enrollment, with blood draws and other evaluations as scheduled. Follow-up assessments will involve weekly app-based questionnaires and a final in-person visit to discuss the study experience, collect weight, and perform a urine drug screen.

ELIGIBILITY:
Example Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced or metastatic solid tumors with any types. This applies to either newly diagnosed cancer or preexisting ones on treatment.
* Patients with active cancers and currently under any line of treatment (please see notable exceptions in the exclusion criteria - patients taking checkpoint inhibitors and investigational agents will not be eligible - also exclusionary medications).
* Patients have been taking their current anti-cancer therapy regimen for at least one month prior to enrollment (to ensure no safety or toxicity issues with study drug initiation).
* Age ≥18 years.
* ECG and lab values demonstrating adequate organ and marrow function at baseline (pre-study).
* Negative urine drug screen for all illicit drugs and THC, CBD prior to randomization
* Ability to understand and the willingness to sign a written informed consent document
* Individuals able to become pregnant will agree to practice an effective form of contraception (e.g., oral birth control pills, condoms, abstinence) for the duration of enrollment (note: urine pregnancy testing will occur monthly)

Exclusion Criteria:

* History of hypersensitivity to cannabis or cannabinoids
* Current, regular use of cannabis/marijuana or THC-containing medications (dronabinol, nabilone) or cannabidiol (Epidiolex) or over-the-counter (OTC) CBD oil.
* Concomitant use of checkpoint inhibitors (e.g., anti-PD1, PDL1, CTLA4) or other drugs for which an cannabinoid interaction may occur.
* Current use of investigational agents, <3 months after the use of investigational agents
* Cardiac conditions contraindicated for cannabis use
* Diagnosis of HPV-related cancer, as there is some evidence that cannabis is contraindicated
* Allergy to any constituent/ingredient contained in the edible dose
* Psychiatric illness/social situations that would limit compliance with study requirements (e.g., bipolar disorder, psychosis, severe depression/anxiety).
* Pregnant or breastfeeding (note: participants will be tested for pregnancy (urine sample) once per month during enrollment)
* Current moderate/severe drug or alcohol use disorder (including cannabis use disorder), positive urine drug screen for illicit drugs or cannabis, or positive alcohol (breathalyzer) during screening
* History of seizure disorder, epilepsy (controlled or uncontrolled)
* Current legal obligations (parole, probation, incarceration, urine drug screen requirements as part of parole/probation/previous incarceration)
* Currently enrolled in substance use treatment
* Self-reported cannabis and synthetic cannabinoid use in the past 30 days (medical or non-medical use is exclusionary)
* Self-reported illicit drug use in past 60 days (ex: methamphetamine, heroin, illicit fentanyl)
* Self-reported daily alcohol use
* Providing a urine sample testing positive for cannabinoids (THC, CBD) or synthetic cannabinoids (K2, Spice-like compounds)
* Providing a sample testing positive for alcohol (breathalyzer) or non-medical use of other drugs (methamphetamine, cocaine) during screening; testing positive during enrollment will lead to discontinuation of the participant's enrollment
* No access to internet/data or devices needed to participate in daily video calls

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2029-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Percent of participants that withdraw from the study or are removed due to adverse events | 5.5 months (includes 2 week no-drug baseline, 4 months of daily dosing, 1 month of no-drug follow-up)
  The percent of patients who elect to withdrawal from the study or removed by physician/investigators due AEs or safety concerns in each group will be measured and compared to the placebo group.

SECONDARY OUTCOMES:
Change in Heart Rate | During each daily dose (daily for 4 months of daily dosing)
  Heart rate data from smart watch gathered immediately prior to and for 4 hours post-dose
Change in O2 saturation | During each daily dose (daily for 4 months of daily dosing)
  O2 saturation data from smart watch gathered immediately prior to and for 4 hours post-dose
Study withdraw rate | 5.5 months (includes 2 week no-drug baseline, 4 months of daily dosing, 1 month of no-drug follow-up)
  Evaluation of the percent of patients who withdraw from the study or removed by physician/investigators for all reasons
Cancer Burden Assessment | 5.5 months (includes 2 week no-drug baseline, 4 months of daily dosing, 1 month of no-drug follow-up)
  Evaluate the effects of cannabis on cancer burden total score Total score will be calculated on a scale of 0-184.

CONTACTS AND LOCATIONS:
Overall Officials: Shanna Babalonis, PhD, Principal Investigator — University of Kentucky College of Medicine; Zin Myint, MD, Principal Investigator — University of Kentucky College of Medicine
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No